CLINICAL TRIAL: NCT01782690
Title: Impact on Survival of Cutaneous Reactions in Erlotinib Plus Gemcitabine Treated Patients With Metastatic Pancreatic Cancer Under Conditions of Daily Routine Practice
Brief Title: An Observational Study of Erlotinib Plus Gemcitabine in Patients With Metastatic Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML23024
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Erlotinib plus Gemcitabine: Patients with metastatic pancreatic cancer, who were planned to receive combination therapy of erlotinib and gemcitabine based on the investigator's assessment.
  Interventions: Drug: erlotinib; Drug: gemcitabine

INTERVENTIONS:
Drug: erlotinib — Study participants will receive erlotinib according to Summary of Product Characteristics (SmPC)
  Other Names: Tarceva
Drug: gemcitabine — Study participants will receive gemcitabine according to Summary of Product Characteristics (SmPC)

SUMMARY:
This observational study will evaluate the impact of rash on survival of patients with metastatic pancreatic cancer treated with erlotinib plus gemcitabine. Further, clinical effectiveness, efficacy and safety will be assessed. Data will be collected for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age >= 18 years
* Patients with metastatic pancreatic cancer where investigators have decided to give combination therapy of erlotinib and gemcitabine according to Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* Contraindications for erlotinib according to Summary of Products Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2012-03-31; Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Klinikum der Universität zu Köln Klinik für Gastroenterologie am Abdominalzentrum, Cologne, Germany

REFERENCES:
- [Derived] Westphalen CB, Kukiolka T, Garlipp B, Hahn L, Fuchs M, Malfertheiner P, Reiser M, Kutting F, Heinemann V, Beringer A, Waldschmidt DT. Correlation of skin rash and overall survival in patients with pancreatic cancer treated with gemcitabine and erlotinib - results from a non-interventional multi-center study. BMC Cancer. 2020 Feb 24;20(1):155. doi: 10.1186/s12885-020-6636-7. PMID 32093649

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib Plus Gemcitabine: Participants with metastatic pancreatic cancer, who were planned to receive combination therapy of erlotinib and gemcitabine based on the investigator's assessment.
Period: Overall Study
Arm/Group | Erlotinib Plus Gemcitabine
Started | 338
Completed | 39
Not Completed | 299
Not completed — Not reported | 7
Not completed — Toxicity of gemcitabine | 1
Not completed — Toxicity of erlotinib | 1
Not completed — Lost to Follow-up | 31
Not completed — Withdrawal of informed consent | 2
Not completed — Absent rash | 9
Not completed — Physician Decision | 13
Not completed — Patient's wish | 21
Not completed — Tumor progression | 74
Not completed — Death | 133
Not completed — Study completion unknown | 7

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all subjects who received at least one treatment with study medication.
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 203

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Stratified by Rash
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause and was stratified by rash status. Participants with rash: rash = yes. Participants without rash: rash = no.
Time Frame: Up to 12 months
Population: Full Analysis Set (FAS) included those enrolled participants who started treatment with erlotinib in combination with gemcitabine.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 270
months
  Rash = Yes | 9.9288 (0.5066) [7.9562 to NA] — N/A=Not Available: Upper Limit not estimable
  Rash = No | 8.6795 (0.3151) [7.2658 to NA] — N/A=Not Available: Upper Limit not estimable
Statistical Analysis 1: Comparison: Erlotinib Plus Gemcitabine; Comparison of Rash=Yes versus Rash=No within Erlotinib plus Gemcitabine arm; Test type: Superiority or Other; p = 0.2361, Log Rank

2. Secondary Outcome: Number of Participants With Rash by Severity
Description: Reported is the total number of participants with rash as well as the number of participants with specific forms of rash, including paronychia, dry skin and papulopustulous eczema. Severity was reported according to Common Terminology Criteria for Adverse Events version 4.0 (CTC AE 4.0): Grade 1 = mild, asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2 = moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily living (ADL); Grade 3 = severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Number; unit: participants
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
participants
  Total number with rash | 174
  Paronychia Grade 1 | 10
  Paronychia Grade 2 | 7
  Paronychia Grade 3 | 2
  Dry skin Grade 1 | 62
  Dry skin Grade 2 | 26
  Papulopustulous eczema Grade 1 | 89
  Papulopustulous eczema Grade 2 | 69
  Papulopustulous eczema Grade 3 | 6

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Number; unit: participants
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
participants | 310

4. Secondary Outcome: Number of Dose Modifications and Dose Withdrawals of Erlotinib
Description: Reported is the total number of dose modifications/withdrawals for erlotinib.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one treatment with study medication
Measure: Number; unit: dose modifications/withdrawals
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
dose modifications/withdrawals | 152

5. Secondary Outcome: Number of Dose Modifications and Dose Withdrawals of Gemcitabine
Description: Reported is the number of dose modifications/withdrawals for gemcitabine.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one treatment with study medication
Measure: Number; unit: dose modifications/withdrawals
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
dose modifications/withdrawals | 738

6. Secondary Outcome: Time of Onset of Rash After Start Erlotinib Treatment
Description: Reported is the number of days from first erlotinib treatment to first rash onset.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
days | 18.4 (21.6)

7. Secondary Outcome: Overall Survival Time Stratified by Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause and was stratified by ECOG-PS at baseline (0-1 versus 2). ECOG-PS 0 = Fully active, able to carry on all pre-disease performance without restriction. ECOG-PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. ECOPG-PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: Up to 12 months
Population: FAS included those enrolled participants who started treatment with erlotinib in combination with gemcitabine.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 270
months
  ECOG-PS grade 0-1 | 9.8301 (0.3726) [8.2192 to NA] — N/A=Not Available: Upper Limit not estimable
  ECOG-PS grade 2 | 6.3452 (0.7396) [4.0110 to NA] — N/A=Not Available: Upper Limit not estimable

8. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response was defined as complete response (CR) plus partial response (PR). Tumor evaluations were performed in accordance with daily routine practice.
Time Frame: Up to 12 months
Population: FAS included those enrolled participants who started treatment with erlotinib in combination with gemcitabine.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 270
percentage of participants | 24.74

9. Secondary Outcome: Time to Disease Progression
Description: Disease progression was defined in accordance with daily routine practice.
Time Frame: Up to 12 months
Population: FAS included those enrolled participants who started treatment with erlotinib in combination with gemcitabine.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 270
months | 4.3726 (0.2945) [3.8795 to 5.0630]

10. Secondary Outcome: Score in Patient Questionnaire: Possible Side Effects
Description: Participant questionnaire regarding satisfaction with the information about possible side effects. Assessment ranged from 1 (very satisfied) to 6 (not satisfied). Questionnaire scores were assessed at several time points during the study.
Time Frame: At Weeks 4, 8, 9 and 16
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
scores on a scale
  Week 4: number analyzed (Participants) | 180
  Week 4 | 1.9 (0.9)
  Week 8: number analyzed (Participants) | 141
  Week 8 | 1.9 (0.9)
  Week 9: number analyzed (Participants) | 1
  Week 9 | 1.0 (NA) — Data based on one participant and therefore standard deviation not available.
  Week 16: number analyzed (Participants) | 94
  Week 16 | 1.9 (0.9)

11. Secondary Outcome: Score in Participant Questionnaire: What to Do in Case of Side Effect
Description: Participant questionnaire regarding satisfaction with the information about what one should do in case of side effects. Assessment ranged from 1 (very satisfied) to 6 (not satisfied). Questionnaire scores were assessed at several time points during the study.
Time Frame: At Weeks 4, 8, 9 and 16
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
scores on a scale
  Week 4: number analyzed (Participants) | 179
  Week 4 | 1.9 (0.8)
  Week 8: number analyzed (Participants) | 140
  Week 8 | 2.0 (1.0)
  Week 9: number analyzed (Participants) | 1
  Week 9 | 1.0 (NA) — Data based on one participant and therefore standard deviation not available.
  Week 16: number analyzed (Participants) | 94
  Week 16 | 1.9 (0.7)

12. Secondary Outcome: Score in Participant Questionnaire: Actual Side Effects of Therapy Compared to Expectation
Description: Participant questionnaire regarding the actual side effects of therapy compared to what one expected before therapy. Assessment ranged from 1 (less than expected) to 6 (more than expected). Questionnaire scores were assessed at several time points during the study.
Time Frame: At Weeks 4, 8, 9 and 16
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
scores on a scale
  Week 4: number analyzed (Participants) | 179
  Week 4 | 2.6 (1.1)
  Week 8: number analyzed (Participants) | 140
  Week 8 | 2.6 (1.1)
  Week 9: number analyzed (Participants) | 1
  Week 9 | 6.0 (NA) — Data based on one participant and therefore standard deviation not available.
  Week 16: number analyzed (Participants) | 94
  Week 16 | 2.7 (1.1)

13. Secondary Outcome: Score in Participant Questionnaire: Quality of Life
Description: Participant assessment of life quality under therapy. Assessment ranged from 1 (very good) to 6 (very bad). Questionnaire scores were assessed at several time points during the study.
Time Frame: At Weeks 4, 8, 9 and 16
Population: Safety population included all participants who received at least one treatment with study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Erlotinib Plus Gemcitabine
Number analyzed (Participants) | 338
scores on a scale
  Week 4: number analyzed (Participants) | 180
  Week 4 | 2.9 (1.1)
  Week 8: number analyzed (Participants) | 140
  Week 8 | 2.9 (1.2)
  Week 9: number analyzed (Participants) | 1
  Week 9 | 1.0 (NA) — Data based on one participant and therefore standard deviation not available.
  Week 16: number analyzed (Participants) | 94
  Week 16 | 2.9 (1.1)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Safety population included all participants who received at least one treatment with study medication.
Arm/Group | Erlotinib Plus Gemcitabine
Serious Adverse Events (participants affected / at risk) | 171/338
Other Adverse Events (participants affected / at risk) | 261/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Plus Gemcitabine (N=338)
Anaemia (Blood and lymphatic system disorders) | 6
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Pyloric stenosis (Congenital, familial and genetic disorders) | 1
Ocular icterus (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Duodenal ulcer (Gastrointestinal disorders) | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastric stenosis (Gastrointestinal disorders) | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 4
Impaired gastric emptying (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Pancreatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Adverse event (General disorders) | 1
Asthenia (General disorders) | 4
Chills (General disorders) | 3
Death (General disorders) | 9
Device dislocation (General disorders) | 2
Device occlusion (General disorders) | 6
Disease progression (General disorders) | 6
Fatigue (General disorders) | 2
General physical health deterioration (General disorders) | 41
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 9
Performance status decreased (General disorders) | 1
Peripheral swelling (General disorders) | 2
Pyrexia (General disorders) | 9
Stent malfunction (General disorders) | 1
Ulcer (General disorders) | 1
Ulcer haemorrhage (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 2
Bile duct stenosis (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 14
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholestatis (Hepatobiliary disorders) | 8
Hepatic failure (Hepatobiliary disorders) | 2
Hydrocholecystis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 8
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cholangitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Endophthalmitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 3
Escherichia infection (Infections and infestations) | 3
Infection (Infections and infestations) | 10
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pulmonary sepsis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Streptococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase abnormal (Investigations) | 1
Blood bilirubin abnormal (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Haemoglobin abnormal (Investigations) | 2
Haemoglobin decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count abnormal (Investigations) | 1
White blood cell count decreased (Investigations) | 2
White blood cell count increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diet refusal (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
IIIrd nerve disorder (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
VIth nerve paralysis (Nervous system disorders) | 1
Disorientation (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Bile duct stent insertion (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 2
Embolism (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Infarction (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
Trousseau's syndrome (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Plus Gemcitabine (N=338)
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 48
Nausea (Gastrointestinal disorders) | 66
Vomiting (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 49
Oedema peripheral (General disorders) | 26
Pain (General disorders) | 61
Infection (Infections and infestations) | 23
Haemoglobin abnormal (Investigations) | 35
Platelet count abnormal (Investigations) | 38
White blood cell count abnormal (Investigations) | 40
Decreased appetite (Metabolism and nutrition disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.